CLINICAL TRIAL: NCT05050942
Title: A Randomized, Multi-center, Open-label, Active-controlled Phase 3 Trial to Assess the Efficacy and Safety of Octreotide Subcutaneous Depot (CAM2029) Versus Octreotide LAR or Lanreotide ATG in Patients With GEP-NET
Brief Title: A Trial to Assess Efficacy and Safety of Octreotide Subcutaneous Depot in Patients With GEP-NET
Acronym: SORENTO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Camurus AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-19-657; 2023-508723-12-00 (EU CTIS Number); 2021-000849-40 (EudraCT Number)
Record Dates: First submitted 2021-09-09; First posted 2021-09-21 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Gastro-enteropancreatic Neuroendocrine Tumor
Keywords: CAM2029; GEP-NET; Octreotide; SORENTO
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAM2029 (Experimental)
  Interventions: Drug: CAM2029
- Octreotide LAR or lanreotide ATG (Active Comparator)
  Interventions: Drug: Octreotide LAR; Drug: Lanreotide ATG

INTERVENTIONS:
Drug: CAM2029 — CAM2029 (octreotide subcutaneous depot) 20 mg will be administered every 2 weeks as a subcutaneous injection
  Arms: CAM2029
Drug: Octreotide LAR — Octreotide LAR 30 mg will be administered every 4 weeks as an intramuscular injection
  Arms: Octreotide LAR or lanreotide ATG
Drug: Lanreotide ATG — Lanreotide ATG 120 mg will be administered every 4 weeks as a deep subcutaneous injection
  Arms: Octreotide LAR or lanreotide ATG

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of CAM2029 to octreotide LAR or lanreotide ATG in patients with advanced, well-differentiated GEP-NET. Patients who experience progressive disease in the randomized part of the study may proceed to an open-label extension part with intensified treatment with CAM2029.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient ≥18 years old
* Histologically confirmed, advanced (unresectable and/or metastatic), and well-differentiated NET of GEP or presumed GEP origin
* At least 1 measurable, somatostatin receptor-positive lesion according to RECIST 1.1 determined by multiphasic CT or MRI (performed within 28 days before randomization)
* ECOG performance status of 0 to 2

Exclusion Criteria:

* Documented evidence of disease progression while on treatment (including SSAs) for locally advanced unresectable or metastatic disease
* Known central nervous system metastases
* Consecutive treatment with long-acting SSAs for more than 6 months before randomization
* Carcinoid symptoms that are refractory to treatment (according to the Investigator's judgement) with conventional doses of octreotide LAR or lanreotide ATG and/or to treatment with daily doses of ≤600 µg of octreotide IR
* Previous treatment with more than 1 cycle of targeted therapies such as mTOR inhibitors or vascular endothelial growth factor inhibitors, or more than 1 cycle of chemotherapy or interferon for GEP-NET
* Treatment of GEP-NET with trans-arterial chemoembolization or trans-arterial embolization within 12 months before screening
* Previously received radioligand therapy (PRRT) at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2021-10-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) as assessed by a Blinded Independent Review Committee (BIRC) | From date of randomization until disease progression or death due to any cause, whichever comes first, assessed up to 48 months
  PFS is defined as time from the date of randomization to the date of the first documented disease progression as per RECIST 1.1 or death due to any cause (whichever occurs first)

SECONDARY OUTCOMES:
Overall survival | Up to 2 years following the primary efficacy analysis
  The time from the date of randomization to the date of death due to any cause
PFS as assessed by local Investigators | From date of randomization until disease progression or death due to any cause, whichever comes first, assessed up to 48 months
  PFS is defined as time from the date of randomization to the date of the first documented disease progression as per RECIST 1.1 or death due to any cause (whichever occurs first)
Overall response rate | From date of randomization until disease progression, assessed up to 48 months
  The proportion of patients with best overall response of complete response (CR) or partial response (PR), as per BIRC according to RECIST 1.1
Disease control rate | From date of randomization until disease progression, assessed up to 48 months
  The proportion of patients with a best overall response of CR, PR or stable disease (SD), as per BIRC according to RECIST 1.1
Time to tumor response | From date of randomization until disease progression, assessed up to 48 months
  The time from the date of randomization to the first documented response of CR or PR, as per BIRC according to RECIST 1.1
Duration of response | From date of randomization until disease progression or death due to underlying cancer, whichever comes first, assessed up to 48 months
  The time from the date of the first documented response of CR or PR to the date of the first documented progression or death due to underlying cancer, as per BIRC according to RECIST 1.1
Incidence of treatment-emergent adverse events | From screening to the safety follow-up, assessed up to 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Simron Singh, MD, MPH, Principal Investigator — Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
Locations (98):
- United States (19):
  - Mayo Clinic Cancer Center (MCCC) - Phoenix, Phoenix, Arizona
  - UCLA Ahmanson Biological Imaging Center, Santa Monica, California
  - Rocky Mountain Cancer Centers - Denver - Midtown, Denver, Colorado
  - Mayo Clinic Hospital - Florida, Jacksonville, Florida
  - Anderson Family Cancer Institute, Jupiter, Florida
  - University of Kentucky (UK) - Markey Cancer Center, Lexington, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The Mount Sinai Hospital, The Bronx, New York
  - White Plains Hospital - Center for Cancer Care, White Plains, New York
  - Texas Oncology - Austin, Austin, Texas
  - Texas Oncology - Dallas, Dallas, Texas
  - Texas Oncology - Denton North, Denton, Texas
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - San Antonio Northeast, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Australia (5):
  - The Queen Elizabeth Hospital (TQEH), Adelaide
  - GenesisCare - North Shore, Alexandria
  - Blacktown Hospital, Blacktown
  - Peter MacCallum Cancer Centre, Melbourne
  - Fiona Stanley Hospital, Murdoch
- Belgium (6):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Hôpital Erasme, Brussels
  - Antwerp University Hospital, Edegem
  - Algemeen Ziekenhuis Maria Middelares, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - AZ Nikolaas, Sint-Niklaas
- Canada (8):
  - London Health Sciences Centre, London
  - Centre Hospitalier de l'Universite de Montreal - Notre-Dame Hospital, Montreal
  - Jewish General Hospital, Montreal
  - The Ottawa Hospital - General Campus, Ottawa
  - Niagara Health System - St. Catharines General Site, St. Catharines
  - Princess Margaret Cancer Centre, Toronto
  - Sunnybrook Health Sciences Centre, Toronto
  - BC Cancer Agency Vancouver Centre, Vancouver
- France (8):
  - CHU Hopitaux de Bordeaux - Hôpital Haut-Lévêque, Bordeaux
  - CHRU de Tours - Hopital Trousseau, Chambray-lès-Tours
  - Centre Hospitalier Universitaire Dijon Bourgogne - L'Hopital General, Dijon
  - Groupe Hospitalier de l'Institut Catholique de Lille - Hopital Saint Vincent de Paul, Lille
  - CHU de Lyon - Groupement Hospitalier Edouard Herriot, Lyon
  - CHU de Nantes - Hôtel-Dieu, Nantes
  - Centre Eugène Marquis, Rennes
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
- Germany (8):
  - Charite - UB - CVK - Medizinische Klinik, Berlin
  - Universitaetsklinikum Erlangen - Hautklinik, Erlangen
  - Universitätsklinikum Essen, Essen
  - Asklepios Klinik St. Georg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Nationales Centrum für Tumorerkrankungen (NCT) Heidelberg, Heidelberg
  - Medizinischen Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Universitätsklinikum Ulm, Ulm
- Hungary (4):
  - SE ÁOK I. sz. Belgyógyászati Klinika, Budapest
  - Petz Aladár Megyei Oktató Kórház, Győr
  - Bács-Kiskun Megyei Kórház, Kecskemét
  - Szegedi Tudományegyetem; I.Belgyógyászati Klinika, Szeged
- Israel (4):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center (HMC) - Hadassah University Hospital (HUH) - Ein Kerem, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (13):
  - Centro di Riferimento Oncologico (CRO), Aviano
  - Universita degli Studi di Bari - Aldo Moro, Bari
  - Azienda Ospedaliero - Universitaria di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - ASST degli Spedali Civili di Brescia, Brescia
  - Universita degli Studi di Firenze - Azienda Ospedaliero - Universitaria Careggi - SC di Oncologia Medical, Florence
  - Universita Degli Studi di Genova - Center of Excellence for Biomedical Research (CEBR), Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori - IRST IRCCS, Meldola
  - Istituto Clinico Humanitas, Milan
  - Azienda Ospedaliero - Universitaria di Modena Policlinico, Modena
  - IRCCS - Istituto Nazionale dei Tumori di Napoli Fondazione G. Pascale - Oncologia Addominale, Napoli
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Azienda Ospedaliera Sant'Andrea, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Trento, Verona
- Netherlands (4):
  - Nederlands Kanker Instituut - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Rijnstate Ziekenhuis - Arnhem, Arnhem
  - Maastricht UMC+, Maastricht
  - Erasmus MC, Rotterdam
- Romania (4):
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuţă" Cluj Napoca, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
  - Sigmedical Services S.R.L., Suceava
- Spain (15):
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall d'Hebron - Vall d'Hebron Institut d'Oncologia (VHIO), Barcelona
  - Institut Catala d'Oncologia Hospitalet, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Facultad de Medicina - Hospital Universitario Fundacion Jimenez Diaz (UAM-FJD) (Clinica de la Concepcion), Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario La Paz (HULP), Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - MD Anderson Cancer Center - Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Parc Taulí Sabadell Hospital Universitari, Sabadell
  - Hospital Universitario Marques de Valdecilla (HUMV), Santander

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh S, Ferone D, Capdevila J, Chan JA, de Herder WW, Halperin D, Mailman J, Hellstrom L, Liedman H, Svedberg A, Tiberg F. Methodology of the SORENTO clinical trial: a prospective, randomised, active-controlled phase 3 trial assessing the efficacy and safety of high exposure octreotide subcutaneous depot (CAM2029) in patients with GEP-NET. Trials. 2024 Jan 16;25(1):58. doi: 10.1186/s13063-023-07834-8. PMID 38229199